CLINICAL TRIAL: NCT06264661
Title: Effect of Cognitive Behavioral Therapy and Phototherapy on Glycosylated Hemoglobin, CLOCK Genes and Quality of Life in Patients With Type 2 Diabetes Mellitus and Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Interdisciplinario de Ciencias de la Salud Unidad Santo Tomás (Other)
Responsible Party: Principal Investigator, Nadia Mabel Pérez Vielma, professor and researcher, Centro Interdisciplinario de Ciencias de la Salud Unidad Santo Tomás
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HJM 006/22-R
Record Dates: First submitted 2024-01-22; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Phototherapy; Glycated Hemoglobin; Quality of Life

STUDY DESIGN:
Intervention Model Description: Clinical, quasi-experimental, pre-post, explanatory, non-probability sampling. Subjects were invited to participate in Hospital Juárez de México. They received eight sessions of Cognitive Behavioral Therapy in combination with phototherapy. The assessment was carried outwith validated instruments for Mexican population and gene expression was evaluated by real-time PCR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Effect of Cognitive Behavioral Therapy with Phototherapy in glycated hemoglobin, CLOCK genes and quality of life in patients with type 2 diabetes mellitus and insomnia — Clinical, quasi-experimental, pre-post, explanatory, non-probability sampling. Subjects were invited to participate in Hospital Juárez de México. They received eight sessions of Cognitive Behavioral Therapy in combination with phototherapy. The assessment was carried out with validated instruments for Mexican population and gene expression was evaluated by real-time PCR.

SUMMARY:
Purpose: To analyze the efficiency of Cognitive Behavioral Intervention in combination with phototherapy to reduce insomnia and improve glycemic control, quality of life, and CLOCK genes expression in patients with type 2 diabetes mellitus. Methods: Clinical, quasi-experimental, pre-post, explanatory, non-probability sampling. Subjects were invited to participate in Hospital Juárez de México. They received eight sessions of Cognitive Behavioral Therapy in combination with phototherapy. The assessment was carried out with validated instruments for Mexican population and gene expression was evaluated by real-time PCR.

ELIGIBILITY:
Inclusion Criteria:

Have a medical record in the Endocrinology service at the Hospital Juarez de Mexico

* Patients with type 2 diabetes mellitus
* Age between 40 and 60 years
* Present Insomnia based on the criteria of The Diagnostic and Diagnostic Manual Statistics of Mental Disorders (DSM-V) which defines insomnia such as predominant dissatisfaction with the quantity or quality of sleep, associated with one (or more) of the following symptoms: a) Difficulty starting the dream,or b) Difficulty maintaining sleep, characterized by awakenings frequent and c) Waking up early in the morning with inability to return to sleep; with clinically significant distress or social impairment, work, educational, academic, behavioral or other important areas of operation, at least three nights a week, for a minimum of three months even with favorable sleeping conditions.
* Sign an informed consent letter and agree to participate in the study.
* Accept taking a blood sample pre and post intervention
* HbA1c level above 6.1% (120 mg/dL;7 mmol/L) or BMI less than 34.9 units

Exclusion Criteria:

* Do not agree to sign the informed consent
* Have a previous psychiatric diagnosis
* Have neurological disorders
* Be diagnosed with type 1 diabetes mellitus or BMI greater than 35 units
* Missing more than 20% of the sessions (2 sessions)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 0 and 3 months
  Pittsburg sleep quality questionnaire,It provides a global rating in 7 components, in no problem, good quality, poor quality and very poor quality of sleep, it consists of 19 multiple option items.
Glycosylated hemoglobin | 0 and 3 months
  A venous blood sample will be taken and analyzed in the clinical analysis laboratory.
Quality of life | 0 and 3 months
  Quality of life questionnaire D39, contains 39 closed items that are grouped into five sections: Energy-Mobility (15 items: 3, 7, 9, 10, 11, 12, 13, 16, 25, 29, 32, 33, 34, 35 and 36), Diabetes control (12 items: 1, 4, 5, 14, 15, 17, 18, 24, 27, 28, 31 and 39); Anxiety-worry (four items: 2, 6, 8 and 22), Social burden (five items: 19, 20, 26, 37 and 38) and Sexual functioning (three items: 21, 23 and 30)
Insomnia | 0 and 3 months
  The Insomnia Scale Athens is made up of eight items, with a scale of Likert type with four response options that ranges of 0 (no sleep-related problem) to 3 (high presence of sleep problems). The first five items identify insomnia and the last three are aimed at identifying consequences of insomnia to the next day

SECONDARY OUTCOMES:
Gene expression analysis of CLOCK | 0 and 3 months
  The determination of gene expression is carried out through the Trizol technique and real-time Polymerase Chain Reaction (PCR-RT) in a 4 ml blood sample taken in tubes with EDTA.
Gene expression analysis of BMAL1 | 0 and 3 months
  The determination of gene expression is carried out through the Trizol technique and real-time Polymerase Chain Reaction (PCR-RT) in a 4 ml blood sample taken in tubes with EDTA.
Gene expression analysis of PER1 | 0 and 3 months
  The determination of gene expression is carried out through the Trizol technique and real-time Polymerase Chain Reaction (PCR-RT) in a 4 ml blood sample taken in tubes with EDTA.
Gene expression analysis of PER2 | 0 and 3 months
  The determination of gene expression is carried out through the Trizol technique and real-time Polymerase Chain Reaction (PCR-RT) in a 4 ml blood sample taken in tubes with EDTA.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Interdisciplinario de Ciencias de la Salud Unidad Santo Tomás, Mexico City, Mexico City, Mexico